CLINICAL TRIAL: NCT06717867
Title: A Randomised, Double-blind Placebo-controlled Study in Healthy Adults to Assess Long Term Population Exposure to Palmitoylethanolamide (Levagen™) to Assess Clinical Safety.
Brief Title: Long-Term PEA Safety Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Collaborators: Gencor Pacific Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: LEVESS
Record Dates: First submitted 2024-11-21; First posted 2024-12-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Safety
Keywords: Palmitoylethanolamide; PEA; Levagen; PEA Safety study
MeSH Terms: interventions — palmidrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEA (Levagen) (Experimental): 600mg PEA each day. 1 oral capsule is taken twice per day after food, each capsule contains 300mg.
  Interventions: Dietary Supplement: Palmitoylethanolamide (PEA)
- Placebo (Placebo Comparator): 600mg microcrystalline cellulose a day. 1 oral capsule is taken twice per day after food, each capsule contains 300mg.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Palmitoylethanolamide (PEA) — Levagen™ capsule containing 300mg Palmitoylethanolamide (PEA). 600mg PEA per day.
  Other Names: Levagen™
  Arms: PEA (Levagen)
Other: Placebo — Placebo capsules contain 300 mg microcrystalline cellulose (MCC), 600mg per day.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn about the long term safety of PEA supplementation in healthy adults. This clinical trial will be in both males and females who are 18 years or older and are healthy volunteers.

The main aim of the study is to assess the safety of long-term use of PEA by assessing the difference between the two groups for serious adverse events, non-serious adverse events, vital signs and biochemistry following 12 months of PEA supplementation.

Participants will:

* Have their suitability for the study checked against the full inclusion/exclusion criteria during the screening process.
* Eligible participants will then complete a baseline visit where assessments will be performed and the participant will be randomly assigned to receive the study product or a placebo. Participants will then consume their assigned study product every day for 12 months. Participants will not know what product they have been assigned during the study.
* Following the baseline visit, there will be 4 visits over 12 months. On months where participants do not have a visit there will be a check in phone call.
* During visits there will be safety assessments performed, blood sampling and questionnaires.

The trial will include two participation modes:

1. In-clinic participation (Brisbane): Participants will attend all visits in-person at the RDC Clinical facility.
2. Remote participation for participants outside of Brisbane: A subgroup of up to 120 participants will participate remotely with virtual visits and at-home assessments. Participants will attend their local pathology centre for blood sampling.

DETAILED DESCRIPTION:
This is an interventional, phase II, randomised, double-blind, placebo-controlled, parallel dose safety study in healthy adults to assess long term population exposure to Palmitoylethanolamide (Levagen™).

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and older)
* Generally healthy
* Able to provide informed consent
* BMI 18.5 - 35.0 kg/m2
* Agree to not participate in another clinical trial during enrolment period

Exclusion Criteria:

* Current malignancy (excluding Basal Cell Carcinoma) or chemotherapy or radiotherapy treatment for malignancy within the previous 2 years
* Serious illness e.g., mood disorders (such as depression or bipolar disorder), anxiety, neurological disorders (such as MS), kidney disease, liver disease or heart conditions
* Unstable illness (e.g., diabetes and thyroid gland dysfunction)
* History of renal function impairment
* Currently taking Coumadin (Warfarin), Heparin, Dalteparin, Enoxaparin or other anticoagulation therapy [(excluding low dose aspirin (under 300 mg/day)]
* Regular consumption (>4 times a week) of PEA over the past 2 weeks
* Substance Abuse (illicit and/or prescription) Drug (prescription or illegal substances) abuse
* Chronic past (within 12-months) and/or current alcohol use (>14 alcoholic drinks week)
* Pregnant or lactating women
* Allergic, sensitive, or intolerant to any of the ingredients in active or placebo formula
* Has a clinically significant abnormal finding on the medical assessment, medical history, or clinical laboratory results at screening.
* Participants who are currently participating in any other clinical trial or who have participated in any other clinical trial during the past 1 month.
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and Female cisgender
Enrollment: 200 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to the end of the study period in participants with SAEs | From Day O (Baseline) to 54 weeks
  Change from baseline to the end of the study period in:
  Number of participants with Serious Adverse Events (SAE) after first administration of study drug through to the last dose of study drug plus 2 weeks [time frame: after first administration of study drug through to the last dose of study drug (12 months) plus 2 weeks (week 54)]

SECONDARY OUTCOMES:
Change from baseline to month 12 in AEs | Baseline (Day 0) to month 12.
  Change from baseline (Day 0, Visit 1) to the end of the study period (month 12, Visit 6) in all adverse events (AEs)
Change from baseline to month 12 in medical assessment | Baseline (day 0) and Month 12
  Change from baseline (Day 0, Visit 1) to the end of the study period (month 12, Visit 6) in safety monitored by Medical assessment (by a doctor).
  The Medical Assessment is a medical review to elucidate symptoms of any occult medical conditions will be conducted for all participants and a medical assessment will then be performed. The assessment will include a review of vital signs and measurements, general appearance, brief cranial nerve assessment, cardiovascular, gastrointestinal and respiratory assessments. Other body systems will be examined (e.g. neurological, renal, musculoskeletal, ear, nose and throat or skin) as is deemed necessary by the trial doctor as guided by the medical review.
Change from baseline to month 12 in Vital Signs (blood pressure) | Baseline (Day 0) to month 12.
  Change from baseline (Day 0, Visit 1) to the end of the study period (month 12, Visit 6) in safety monitored by blood pressure (mmHg).
Change from baseline to month 12 in Vital Signs (heart rate) | Baseline (Day 0) to month 12.
  Change from baseline (Day 0, Visit 1) to the end of the study period (month 12, Visit 6) in safety monitored by heart rate (bpm).
Change from baseline to month 12 in clinical laboratory determinations (Full Blood Count) | Baseline (Day 0) to month 12.
  Change from baseline (Day 0, Visit 1) to the end of the study period (month 12, Visit 6) in safety monitored by Full Blood Count (FBC).
Change from baseline to month 12 in clinical laboratory determinations (fasting glucose) | Baseline (Day 0) to month 12.
  Change from baseline (Day 0, Visit 1) to the end of the study period (month 12, Visit 6) in safety monitored by fasting glucose.
Change from baseline to month 12 in clinical laboratory determinations (insulin) | Baseline (Day 0) to month 12.
  Change from baseline (Day 0, Visit 1) to the end of the study period (month 12, Visit 6) in safety monitored by insulin.
Change from baseline to month 12 in clinical laboratory determinations (lipids). | Baseline (Day 0) to month 12.
  Change from baseline (Day 0, Visit 1) to the end of the study period (month 12, Visit 6) in safety monitored by lipids.
Change from baseline to month 12 in clinical laboratory determinations (electrolytes) | Baseline (Day 0) to month 12.
  Change from baseline (Day 0, Visit 1) to the end of the study period (month 12, Visit 6) in safety monitored by electrolytes.
Change from baseline to month 12 in clinical laboratory determinations (kidney function tests) | Baseline (Day 0) to month 12.
  Change from baseline (Day 0, Visit 1) to the end of the study period (month 12, Visit 6) in safety monitored by kidney function tests.
Change from baseline to month 12 in clinical laboratory determinations (Liver function tests) | Baseline (Day 0) to month 12.
  Change from baseline (Day 0, Visit 1) to the end of the study period (month 12, Visit 6) in safety monitored by liver function tests.
Change from baseline to month 12 in sleep questionnaires. | Baseline (Day 0) to month 12.
  Change from baseline (Day 0) to the end of the study period (month 12) in safety monitored by Leeds sleep evaluation questionnaire (LSEQ).
  Each domain of the LSEQ is scored using a visual analogue scale (VAS) where participants mark their response on a line ranging from 0 to 100.
  Higher scores indicate better sleep quality or easier sleep-related behaviors in the respective domain. Lower scores indicate poorer sleep quality or more difficulty in the respective domain.
Change from baseline to month 12 in anxiety questionnaires | Baseline (Day 0) to month 12.
  Change from baseline (Day 0) to the end of the study period (month 12) in safety monitored by Anxiety questionnaires (Beck Anxiety Inventory Scale). Scores from 0 to 63, a score of 0-21 indicates low anxiety whereas a score of 36 and above indicates potentially concerning levels of anxiety.
Change from baseline to month 12 in Quality of life | Baseline (Day 0) to month 12.
  Change from baseline (Day 0) to the end of the study period (month 12) in safety monitored by Quality of life (RAND 36-Item Short Form Survey Instrument, Rand SF-36).
Change from baseline to month 12 in Musculoskeletal health questionnaire | Baseline (Day 0) to month 12.
  Change from baseline (Day 0) to the end of the study period (month 12) in safety monitored by Musculoskeletal health questionnaire (MSK-HQ). MSK-HQ is scored on a range of 0-56, with a better score indicating better MSK-HQ health status.
Change from baseline to month 12 in Gastrointestinal tolerance questionnaire | Baseline (Day 0) to month 12.
  Change from baseline (Day 0) to the end of the study period (month 12) in safety monitored by Gastrointestinal tolerance questionnaire

OTHER OUTCOMES:
Exploratory: Change from baseline to month 12 in Vital Signs (temperature) | Baseline (Day 0) to month 12.
  Change from baseline (Day 0, Visit 1) to the end of the study period (month 12, Visit 6) in safety monitored by temperature (celcius).
Exploratory: Change from baseline to month 12 in Vital Signs (O2 saturation) | Baseline (Day 0) to month 12.
  Change from baseline (Day 0, Visit 1) to the end of the study period (month 12, Visit 6) in safety monitored by O2 saturation (%).
Exploratory: Change from baseline to month 12 in PEA | Baseline (Day 0) to month 12.
  Change from baseline (Day 0, Visit 1) to the end of the study period (month 12, Visit 6) in PEA plasma concentration over time
Exploratory: Change from baseline to month 12 in serum BDNF, CRP, and cytokines | Baseline (Day 0) to month 12.
  Change from baseline (Day 0) to the end of the study period (month 12) in safety monitored by Serum BDNF, CRP, and cytokines (e.g., IL-1b, IL-6, IL-10, TNF-a)]

CONTACTS AND LOCATIONS:
Locations (1):
- RDC Clinical, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No